CLINICAL TRIAL: NCT07112404
Title: PINPOINT Study: Pain Intervention With Needling: Pilot Of Integrated Neuromodulation Techniques
Brief Title: Pain Intervention With Needling: Pilot Of Integrated Neuromodulation Techniques
Acronym: PINPOINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-0109; K12NS130673 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-08-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Pain; Back Pain; Lower Back Pain; Quality of Life
MeSH Terms: conditions — Pain; Back Pain; Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry Needling Only Group (Experimental): This group will receive dry needling only. The group will receive the dry needling at visits 2-7.
  Interventions: Other: Dry Needling
- Dry Needling Plus high-rate PENS (Experimental): This grouping will receive dry needling plus high-rate PENS. The group will receive the dry needling at visits 2-7.
  Interventions: Other: Dry needling with high-rate PENS
- Dry Needling Plus low-rate PENS (Experimental): This grouping will receive dry needling plus low-rate PENS. The group will receive the dry needling at visits 2-7.
  Interventions: Other: Dry needling with low-rate PENS

INTERVENTIONS:
Other: Dry Needling — Dry needling is a therapeutic technique where thin, solid filiform needles are inserted into trigger points, tight muscle bands, or areas of muscle tension without injecting any medication. The procedure aims to release muscle knots, reduce pain, and improve muscle function by stimulating the body's natural healing response.
  Arms: Dry Needling Only Group
Other: Dry needling with high-rate PENS — Dry needling is a therapeutic technique where thin, solid filiform needles are inserted into trigger points, tight muscle bands, or areas of muscle tension without injecting any medication. The procedure aims to release muscle knots, reduce pain, and improve muscle function by stimulating the body's natural healing response.
  When combined with high-rate percutaneous electrical nerve stimulation (PENS), the needles serve as electrodes for delivering a controlled, high-frequency electrical current directly to the targeted tissues. This electrical stimulation further modulates pain signals, promotes muscle relaxation, and can enhance the effectiveness of dry needling, especially for persistent pain and neuromuscular dysfunction.
  Arms: Dry Needling Plus high-rate PENS
Other: Dry needling with low-rate PENS — Dry needling is a therapeutic technique where thin, solid filiform needles are inserted into trigger points, tight muscle bands, or areas of muscle tension without injecting any medication. The procedure aims to release muscle knots, reduce pain, and improve muscle function by stimulating the body's natural healing response.
  When combined with low-rate percutaneous electrical nerve stimulation (PENS), the needles serve as electrodes for delivering a controlled, low-frequency electrical current directly to the targeted tissues. This electrical stimulation further modulates pain signals, promotes muscle relaxation, and can enhance the effectiveness of dry needling, especially for persistent pain and neuromuscular dysfunction.
  Arms: Dry Needling Plus low-rate PENS

SUMMARY:
The study's purpose is to determine the effects of three different dry needling sessions on pain and quality of life for those with chronic low back pain. Dry needling is a therapeutic procedure in which a very thin, monofilament needle is inserted through the skin to reach a target tissue like a muscle to help reduce pain, improve muscle activation, and increase blood flow. Dry needling has also been shown to improve nervous system function.

DETAILED DESCRIPTION:
Phase 1: Specific Aim 1 Once IRB approval is granted, the research team will initiate participant recruitment for Phase 1. This phase aims to recruit participants over a period of 4 months or until 12 participants are enrolled. Participants will be asked to wear comfortable clothing that allows them to move easily and allows access to the lumbar region.

Participants will be expected to participate in 3 sessions. Session 1 will last up to 120 minutes (2 hours), session 2 is expected to last up to 1 hour, and session 3 up to 120 minutes (2 hours). Depending on scheduling availability, participants can be expected to be a part of the study for 1 to 2 weeks. Each session will be at least 1 day apart (24 hours) to allow for their health systems to return to baseline.

Upon completion of data collection, the study team will aim to develop a protocol for publication and disseminate other relevant findings.

Phase 2: Specific Aim 2 Recruitment for Phase 2 will begin once the recruitment procedures for Phase 1 are reviewed with a goal of recruiting 30 participants, 10 in each group. Prior to beginning the study, participants will complete the informed consent for phase 2.

Participants will be block-randomized into one of three intervention groups. Participants in the intervention groups will be expected to participate in a baseline assessment, 6 intervention visits, a 2nd assessment, at least 2 weeks of wash out, a post-intervention assessment with a one-on-one interview, and a one- and three-month survey follow-up. Figure 2 outlines the flow of participation. Participants will be asked to wear comfortable clothing that allows them to move easily and allows access to the lumbar region.

Assessments and interventions are anticipated to be completed within 2 months. When including the follow-up surveys, the total time for participants in this phase to be in the study is anticipated to be 4 to 5 months. The proposed work for study 2 is anticipated to be completed in approximately 1 year with an additional 6 months for manuscript development.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females between the ages of 18 and 65 will be included in this study.

Phase 1 Inclusion criteria

- Healthy adults who report no pain for more than 1 day in the past 3 months in their lumbar region. Lumbar region will include posterior lumber musculature, lumbar spine, sacroiliac pain, or superior gluteal area pain.

Phase 2 Inclusion criteria

* Adults experiencing chronic low back pain. Chronic low back pain will be identified as having pain the lumbar region for at least 3 months. The pain may be constant or episodic in nature.
* Participants will be included if they experience pain at least 75% of the days in the past 3 months. All pain levels will be included. Lumbar region will include posterior lumber musculature, lumbar spine, sacroiliac pain, or superior gluteal area pain.

Exclusion Criteria:

* Individuals who are currently seeking any form of medical treatment for lumbar conditions beyond routine physician follow-up appointments in order to avoid confounding variables, regardless of pain-free status. These may include, but are not limited to, seeking treatment from a chiropractor, acupuncturist, or massage therapist or medical procedures such as injections into the lumbar region for pain.
* Additionally, those with previous lumbar surgeries or those with previous major injuries to the lumbar spine that may have resulted in structural abnormalities that may compromise needle placement will be excluded. If surgical procedures did not alter structural alignment, then it will be allowed. For example, an approved procedure may include discectomy or nerve ablation, while a not approved procedure would include a lumbar fusion or scoliosis rod placement.
* Additionally, if a person is experiencing radicular symptoms from a back injury, despite not feeling the symptoms in the lumbar region, will not be considered. Radicular symptoms will be defined as those present past the knee and/or electrical in nature. Individuals with neurological conditions or those who need the services of another due to cognitive deficits will not be considered for this study.
* Furthermore, as this study relies on an intact sensory system, participants with conditions that may affect sensory processing (e.g., peripheral neuropathy, skin conditions, or circulatory disorders) will be excluded through careful screening.

Additional exclusion criteria

* Will include the following conditions identified as contraindications for dry needling: those with impaired sensitivity, taking anticoagulants, a compromised immune system, a local or systemic infection, an active tumor, history of lymph node removal, history of autoimmune disease, allergy to metals such as nickel or chromium, history of cosmetic procedures in the area, pregnant individuals, or osteoporosis.
* Non-English-speaking subjects will be excluded from the study due to the need to understand any communication while dry-needling procedures are taking place.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Assess the acceptability and feasibility of the protocol- Phase 1 Healthy Participants | one week, up to 3 months
  Acceptability and feasibility will be assessed through an interview and retention records at the end of the study.
Assess the acceptability and feasibility of the protocol- Phase 2 Those with Chronic Low Back Pain | 3 months, up to 2 years.
  Acceptability and feasibility will be assessed through an interview and retention records at the end of the study.

SECONDARY OUTCOMES:
Physiological Activity Level Measured by ActiGraph for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  Time spent in sedentary, low-intensity, and moderate-to-vigorous physical activity. Physical activity will be measured while enrolled in the study using the ActiGraph GT9X accelerometers. Higher = More activity (better).
Physiological Activity Level Measured by Shimmer3 Galvanic Skin Response(GSR) +Unit for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  Lower GSR often indicates less arousal.
Physiological Activity Level Measured by Shimmer3 ECG Unit for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  Beats per minute (BPM) will be collected and assessed from baseline while utilizing dry needling procedures.
Physiological Activity Level Measured by Clario Opal for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  Clario Opal-often called the Opal V2C® System-is a medical-grade wearable sensor solution that captures objective digital endpoints of mobility. It tracks gait, balance, and other functional mobility tasks using validated protocols and analytics. Higher gait speed/balance = better.
Michigan Visual Stress Test (M-VAST) for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The Michigan Visual Stress Test (M-VAST) produces a total visual stress symptom score ranging from 0 (no symptoms) to 30 (severe symptoms), based on participant self-reports across 10 visual stress indicators. A higher score indicates greater severity of visual discomfort or distortion.
Physical Assessment Measured by 6-minute walk test for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The 6-Minute Walk Test (6MWT) is a standardized functional performance measure in which participants are instructed to walk for 6 minutes along a marked 30-meter indoor course. The total distance walked (in meters) is recorded. The 6-Minute Walk Test (6MWT) is a standardized functional performance measure in which participants are instructed to walk for 6 minutes along a marked 30-meter indoor course. The total distance walked (in meters) is recorded.
Self-Reported Outcome Measured by Numeric Pain Rating Scale for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The Numeric Pain Rating Scale (NPRS) is a self-reported measure of pain intensity. Participants are asked to rate their pain on an 11-point scale ranging from 0 to 10, where 0 = no pain and 10 = worst pain imaginable. Lower scores indicate lower pain intensity.
Self-Reported Outcome Measured by PROMIS-29+2 for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The PROMIS-29+2 is a standardized self-reported questionnaire that assesses 8 health domains: physical function, anxiety, depression, fatigue, sleep disturbance, social roles, pain interference, and cognitive function. It includes 29 items from the PROMIS-29 plus 2 cognitive function items and a single 0-10 numeric rating for pain intensity. Each domain is scored using T-scores (mean = 50, SD = 10), with higher scores indicating more of the measured concept (e.g., greater fatigue or better physical function, depending on the domain).
Self-Reported Outcome Measured by Roland-Morris Disability Questionnaire for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The Roland-Morris Disability Questionnaire is a 24-item self-reported tool used to assess functional disability due to low back pain. Each item describes a limitation in daily activities related to physical function. Minimum Score: 0 (no disability) Maximum Score: 24 (maximum disability) Higher scores indicate greater disability due to back pain.
Self-Reported Outcome Measured by Patient-Specific Functional Scale for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The Patient-Specific Functional Scale (PSFS) is a validated, individualized tool used to measure a patient's ability to perform activities that are personally important but limited due to injury or condition. Participants identify up to 5 activities limited by their condition and rate their ability to perform each on a scale from 0 (unable) to 10 (same as before problem). The average score across all reported activities is used for analysis. Higher scores reflect better function.
Self-Reported Outcome Measured by Complex Medical Symptoms Inventory for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The CMSI includes 52 items representing somatic symptoms experienced persistently (≥3 months) over the past year or lifetime. Scores range from 0 (no symptoms) to 52 (maximum symptoms), with higher scores reflecting greater multisystem symptom complexity and burden.
Self-Reported Outcome Measured by World Health Organization Quality of Life Instrument for Phase 1 and Phase 2(WHOQOL) | 1 day (30-60 minutes)
  The WHOQOL-BREF is a 26-item self-report instrument developed by the World Health Organization to assess quality of life across four domains: physical health, psychological health, social relationships, and environment. Scores are transformed to a 0-100 scale, with higher scores indicating better quality of life.
Self-Reported Outcome Measured by Tobacco, Alcohol, Prescription Drug, and Illicit Substance Use Tool (TAPS Part 1) for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The TAPS Part 1 Tool is a self-administered or interviewer-administered instrument designed to screen for past-year and past-3-month use of tobacco, alcohol, illicit drugs, and the nonmedical use of prescription medications. Higher scores indicate more frequent use and potential risk for a substance use disorder. Scores range from 0 to 20, higher is better.
Self-Reported Outcome Measured by Patient Global Impression of Change (PGIC) for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The PGIC is a single-item instrument scored from 1 (very much improved) to 7 (very much worse). A lower score reflects greater perceived improvement. Responses of 1 ("very much improved") or 2 ("much improved") are considered indicative of clinically meaningful improvement.
Self-Reported Outcome Measured by Generalized Anxiety Disorder for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The GAD-7 is scored from 0 (no anxiety) to 21 (severe anxiety), with higher scores indicating greater symptom severity. A score ≥10 is suggestive of clinically significant generalized anxiety disorder.
Self-Reported Outcome Measured by Patient Health Questionnaire for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The Patient Health Questionnaire is scored from 0 (no depression) to 27 (severe depression), with higher scores indicating greater symptom severity.
Self-Reported Outcome Measured by Pain Catastrophizing Scale for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The PCS is a 13-item instrument scored from 0 (not at all) to 4 (all the time), with a total score range of 0-52. Higher scores indicate greater pain catastrophizing.
Self-Reported Outcome Measured by Sleep Disturbance for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  PROMIS Sleep Disturbance T-scores range approximately from 20 to 80. Higher scores indicate greater sleep disturbance or poorer sleep quality. Lower scores reflect better or normal sleep.
Self-Reported Outcome Measured by Pain, Enjoyment of Life, and General Activity (PEG) for Phase 1 and Phase 2 | 1 day (30-60 minutes)
  The PEG is a 3-item scale scored from 0 (no pain/interference) to 10 (worst pain/completely interferes). The total score is the mean of the three items, with higher scores indicating greater pain severity and impact.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Medical Branch, Galveston, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No